CLINICAL TRIAL: NCT02324231
Title: SPOG 2015 FN Definition. A Swiss Pediatric Oncology Group (SPOG) Initiated Multi-center Open-label Randomized Controlled Multiple Crossover Non-inferiority Trial on Safety of a High Versus Low Temperature Limit Defining Fever in Pediatric Patients With Cancer at Risk for Fever in Chemotherapy-induced Neutropenia (FN)
Brief Title: SPOG 2015 FN Definition. A Multi-center Non-inferiority Trial on Safety of a High Versus Low Temperature Limit Defining Fever in Pediatric Patients With Cancer at Risk for Fever in Chemotherapy-induced Neutropenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Pediatric Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SPOG 2015 FN Definition
Record Dates: First submitted 2014-12-18; First posted 2014-12-24 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2018-10

CONDITIONS: Cancer; Pediatrics; Fever; Neutropenia; Fever in Neutropenia
MeSH Terms: conditions — Neoplasms; Fever; Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 39.0°C temperature limit defining fever (Other): Temperature limit defining fever, for definition of fever in neutropenia (FN), is single temperature >=39.0°C measured in the ear by infrared tympanic thermometry. If clinically indicated, the treating physician is allowed to make the diagnosis of FN at lower temperatures.
  Interventions: Other: 39.0°C temperature limit defining fever
- 38.5°C temperature limit defining fever (Other): Temperature limit defining fever, for definition of fever in neutropenia (FN), is single temperature >=38.5°C measured in the ear by infrared tympanic thermometry. If clinically indicated, the treating physician is allowed to make the diagnosis of FN at lower temperatures.
  Interventions: Other: 38.5°C temperature limit defining fever

INTERVENTIONS:
Other: 39.0°C temperature limit defining fever — Diagnosis of FN, correspondingly hospitalization and start of empirical intravenous broad-spectrum antimicrobial therapy. Further treatment according to treating physician.
  Arms: 39.0°C temperature limit defining fever
Other: 38.5°C temperature limit defining fever — Diagnosis of FN, correspondingly hospitalization and start of empirical intravenous broad-spectrum antimicrobial therapy. Further treatment according to treating physician.
  Arms: 38.5°C temperature limit defining fever

SUMMARY:
In a multi-center open-label cluster-randomized controlled parallel-group multiple crossover non-inferiority trial in children and adolescents up to 20 years diagnosed with cancer requiring chemotherapy, primarily the safety, and secondarily the efficacy and other endpoints, of a high (39.0°C) versus low (38.5°C) temperature limit defining fever (TLDF) for the diagnosis of fever in chemotherapy-induced neutropenia (FN) is studied. Safety is assessed by the rate of safety relevant events per chemotherapy exposure time, a composite endpoint including serious medical complications and bacteremia during FN. Patients are repeatedly randomized (cluster: study site) to the high or the low TLDF every month, resulting in possible multiple crossovers in one patient. The high TLDF is declared not to be inferior regarding safety compared to the low TLDF if non-inferiority of the rate ratio of safety relevant events is proven, with a single-sided non-inferiority margin of 1.33, applying mixed Poisson regression.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy treatment because of any malignancy for at least 2 months at time of recruitment for myelosuppressive therapy, or at least 1 cycle of myeloablative chemotherapy followed by autologous hematopoietic stem cell transplantation
* Age ≥12 months and <18 years at time of recruitment
* Written informed consent from patients and/or parents

Exclusion Criteria:

* Infants <1 years old (reason: differences in temperature measurement method)
* Past allogeneic hematopoietic stem cell transplantation
* Denied written informed consent from patients and/or parents

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 269 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Rate of clinically defined FN with at least one safety relevant event | 1 year (estimated average)
  Poisson rate: number of clinically defined FN with at least one SRE divided by the entire chemotherapy exposure time for each patient, estimated to be 1 year on average (Unit: FN per year of chemotherapy exposure time) SRE: Composite endpoint (serious medical complication AND/OR bacteremia), reached until the end of each individual FN episode (Unit: binary)

SECONDARY OUTCOMES:
Times and delays of diagnosis and therapy (A) | 1 year (estimated average)
  Times (hh:mm) of measurement of fever - telephone to study site - arrival at emergency department - prescription of antibiotics - start and end of first dose of i.v. antibiotics (assessed per FN episode by the responsible local PHO and in patient chart, reported per FN episode; unit: hours:minutes)
Adverse events (B) | 1 year (estimated average)
  AE: clinically / microbiologically documented infection, unexplained fever, sepsis / severe sepsis / septic shock, relapse of primary infection (assessed in patient charts, reported per FN; unit:binary)
Delay from crossing low to high TLDF (C) | 1 year (estimated average)
  Only for currently active high TLDF: delay time between crossing low and high TLDF; delayed FN diagnosis (see 5.1.4) by high vs. low TLDF (assessed from patients charts, reported per FN; unit: hours:minutes)
Rate of clinically defined FN (D) | 1 year (estimated average)
  Poisson rate: number of clinically defined FN divided by the entire chemotherapy exposure time for each patient, estimated to be 1 year on average (Unit: FN per year of chemotherapy exposure time)
Rate of FN diagnosed at/above TLDF (E) | 1 year (estimated average)
  Poisson rate: number of FN diagnosed at/above TLDF divided by the entire chemotherapy exposure time for each patient, estimated to be 1 year on average (Unit: FN per year of chemotherapy exposure time)
Rate of FN diagnosed below TLDF (E) | 1 year (estimated average)
  Poisson rate: number of FN diagnosed below TLDF divided by the entire chemotherapy exposure time for each patient, estimated to be 1 year on average (Unit: FN per year of chemotherapy exposure time)
Duration of treatment (F) | 1 year (estimated average)
  . Duration of hospitalization, ICU treatment, i.v. antibiotics, p.o. antibiotics, any antibiotics, delay of chemotherapy for FN (unit: days)
Simultaneous and avoided FN diagnoses (G) | 1 year (estimated average)
  Only for currently active high TLDF: Simultaneous and avoided FN diagnoses by high vs. low TLDF (assessed from patients charts, reported per FN; unit: binary)

OTHER OUTCOMES:
Development of rules predicting risk of FN during chemotherapy | 1 year (estimated average)
  Risk prediction rules for clinically defined FN, clinically defined FN with bacteremia, with serious medical complication, and with safety relevant event during chemotherapy, all based on multivariate mixed Poisson regression (stepwise forward variable selection procedure; unit: predictor)
Development of rules predicting risk of adverse events during FN | 1 year (estimated average)
  Risk prediction rules for bacteremia, for serious medical complication, and for safety relevant event during FN, all based on multivariate mixed logistic regression (stepwise forward variable selection procedure; unit: predictor)
External validation of rules predicting risk of FN during chemotherapy | 1 year (estimated average)
  Validation of published risk prediction rules for clinically defined FN, clinically defined FN with bacteremia, with serious medical complication, and with safety relevant event during chemotherapy (units: sensitivity, specificity, positive and negative predictive value, area under receiver operating characteristic curve)
External validation of rules predicting risk of adverse events during FN | 1 year (estimated average)
  Validation of published risk prediction rules for bacteremia, for serious medical complication, and for safety relevant event during FN (units: sensitivity, specificity, positive and negative predictive value, area under receiver operating characteristic curve)

CONTACTS AND LOCATIONS:
Overall Officials: Roland A Ammann, MD, Study Chair — Universitätsklinik für Kinderheilkunde, Inselspital, Bern
Locations (6):
- Switzerland (6):
  - Basel: Universitätskinderklinik beider Basel, Basel
  - Bern: Universitätsklinik für Kinderheilkunde, Inselspital, Bern
  - Geneva: Département de Pédiatrie, Hôpital Cantonal de Genève, Geneva
  - Lausanne: Hémato-Oncologie Pédiatrique, CHUV, Lausanne
  - Luzern: Pädiatrische Hämatologie/Onkologie, Kinderspital, Lucerne
  - Zürich: Pädiatrische Onkologie Kinderspital, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ammann RA. A sequence of Swiss studies on the temperature Limit defining fever in pediatric oncology. Schweizer Krebsbulletin 35(1): 69-71, 2015.
- [Derived] Lavieri L, Koenig C, Bodmer N, Agyeman PKA, Scheinemann K, Ansari M, Roessler J, Ammann RA. Predicting fever in neutropenia with safety-relevant events in children undergoing chemotherapy for cancer: The prospective multicenter SPOG 2015 FN Definition Study. Pediatr Blood Cancer. 2021 Dec;68(12):e29253. doi: 10.1002/pbc.29253. Epub 2021 Jul 26. PMID 34310027
- [Derived] Koenig C, Bodmer N, Agyeman PKA, Niggli F, Adam C, Ansari M, Eisenreich B, Keller N, Leibundgut K, Nadal D, Roessler J, Scheinemann K, Simon A, Teuffel O, von der Weid NX, Zeller M, Zimmermann K, Ammann RA. 39.0 degrees C versus 38.5 degrees C ear temperature as fever limit in children with neutropenia undergoing chemotherapy for cancer: a multicentre, cluster-randomised, multiple-crossover, non-inferiority trial. Lancet Child Adolesc Health. 2020 Jul;4(7):495-502. doi: 10.1016/S2352-4642(20)30092-4. Epub 2020 Jun 1. PMID 32497520

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT02324231/Prot_SAP_000.pdf